CLINICAL TRIAL: NCT02913716
Title: A Phase I, Open-label Study of the Absorption, Metabolism and Excretion of Defactinib (VS-6063-106) in Healthy Male Subjects
Brief Title: A Phase I, Open-label Study of Absorption, Metabolism, and Excretion of Defactinib (VS-6063) in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VS-6063-106
Record Dates: First submitted 2016-09-19; First posted 2016-09-26 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — defactinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Defactinib treatment (Experimental): Single dose of 400 mg [14C]-defactinib, oral suspension
  Interventions: Drug: defactinib

INTERVENTIONS:
Drug: defactinib — Single oral dose of 400 mg [14C]-defactinib
  Other Names: VS-6063

SUMMARY:
This study assesses the mass balance recovery, pharmacokinetics, metabolite profile and metabolite identification of defactinib.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 18.0 to 35.0 kg/m2
* History (Hx) regular bowel movements
* Creatinine clearance >80 mL/min

Exclusion Criteria:

* Hx alcohol abuse in past 2 yrs
* Current smoker
* Systolic blood pressure (S) or diastolic blood pressure (DBP) above upper limit of reference range (age 40-44 >90/140; age 45-65 >90/150)

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Urine amount excreted (Ae) | Screening to 168h post-dose
Urine fraction of the dose excreted (Fe) | Screening to 168h post-dose
Urine cumulative amount excreted (Cum Ae) | Screening to 168h post-dose
Urine cumulative fraction of the dose excreted (Cum Fe) | Screening to 168h post-dose
Urine renal clearance (CLr) | Screening to 168h post-dose
Faeces Ae | Screening to 168h post-dose
Faeces Fe | Screening to 168h post-dose
Faeces Cum Ae | Screening to 168h post-dose
Faeces Cum Fe | Screening to 168h post-dose
All excreta Ae | Screening to 168h post-dose
All excreta Fe | Screening to 168h post-dose
All excreta Cum Ae | Screening to 168h post-dose
All excreta Cum Fe | Screening to 168h post-dose
All excreta non-renal clearance (CLnr) | Screening to 168h post-dose

SECONDARY OUTCOMES:
Time at which the analyte is first quantifiable (Tlag) | Screening to 168h post-dose
Time from dosing at which Cmax is apparent (Tmax) | Screening to 168h post-dose
Maximum observed concentration (Cmax) | Screening to 168h post-dose
Area under the concentration vs. time curve from time zero extrapolated to last measurable concentration (AUC(0-last)) | Screening to 168h post-dose
Area under the concentration vs. time curve from time zero to infinity (AUC (0-inf)) | Screening to 168h post-dose
Percentage of AUC(0-inf) accounted for by extrapolation (AUC%extrap) | Screening to 168h post-dose
lamdba-z | Screening to 168h post-dose
Apparent elimination half-life (T1/2) | Screening to 168h post-dose
Mean residence time | Screening to 168h post-dose
Apparent clearance after oral administration (CL/F) | Screening to 168h post-dose
Apparent volume of distribution after oral administration (Vz/F) | Screening to 168h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, Study Chair — Verastem, Inc.

IPD SHARING:
Plan to Share IPD: No